CLINICAL TRIAL: NCT06730217
Title: Bronchial Clearance Carried Out With a Mechanical In-exsufflator vs. a Manual Respiratory Physiotherapy Technique in Hospitalized Elderly People
Acronym: INEXPA2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RBHP 2024 ESTENNE; 2024-A01839-38 (Other: 2024-A01839-38)
Record Dates: First submitted 2024-11-29; First posted 2024-12-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-11

CONDITIONS: Bronchial Congestion; Airway Clearance Impairment
Keywords: respiratory muscle; mechanical ventilators; bronchial congestion
MeSH Terms: interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Participants randomized to the intervention group will benefit from a mechanical insufflator during airway clearance sessions (EOVE-70®, Air Liquide Medical Systems France). In this group, patients will also be assessed before and after each session, in order to compare the 2 chosen airway clearance techniques on variation in peak expiratory flow.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants randomized to the control group will receive standard care. The patient is then assessed by a first physiotherapist evaluator, who measures the data described in the study setting section. The physiotherapist then performs a manual bronchial decongestion session, using the Expiratory Flow Augmentation technique with abdominal and thoracic counter-pressure.
  Interventions: Other: Control : standard care
- Experimental (Experimental): Participants randomized to the intervention group will benefit from a mechanical insufflator during airway clearance sessions (EOVE-70®, Air Liquide Medical Systems France).
  Interventions: Device: Intervention : mechanical insufflator

INTERVENTIONS:
Device: Intervention : mechanical insufflator — Participants randomized to the intervention group will benefit from a mechanical insufflator during airway clearance sessions (EOVE-70®, Air Liquide Medical Systems France).
  Other Names: Device
  Arms: Experimental
Other: Control : standard care — Participants randomized to the control group will receive standard care
  Arms: Control

SUMMARY:
Everywhere in the world, life expectancy is increasing. Currently, most individuals can expect to live up to 60 years and beyond. In all countries, the number and proportion of older adult in the population are rising. By 2030, one in six people in the world will be 60 years old or older.

France is also seeing its population age, with the number of older people increasing from 14% in 2014 to 21% in 2022. In 2018, elderly people accounted for 30% of short-stay hospitalizations. One of the most common causes of hospitalization for older adult is respiratory system pathologies, second only to cardiovascular system pathologies. Admission for a respiratory pathology is often associated with bronchial congestion. Infectious or viral pneumonia is often the terminal illness for the older adult. In the United States, 1 million old patients are hospitalized for this pathology, and 30% of them will die within the year.

Old people are more susceptible to pneumonia due to several factors, including impaired gag reflex, reduced muco-ciliary function, weakened immunity, impaired fever response, and various degrees of cardiopulmonary dysfunction. Additionally, central nervous system disorders and/or impaired gag reflex increase the risk of aspiration pneumonia in old patients. The majority of these patients develop a productive cough, but unfortunately, their ability to cough effectively is often reduced.

Aging leads to various changes in the respiratory system. The thoracic cage and spine deform due to calcification and osteoporosis, resulting in stiffness. The thoracic wall stiffens, making mobilization more difficult and increasing the muscular work required for expansion during inspiration. The diaphragm is in a less favorable position to contract effectively. Expiration becomes less efficient, leading to an increase in residual volume (RV) and promoting what is called "senile emphysema," where air spaces dilate and dead spaces increase. This leads to an increase in functional residual capacity and RV, reducing vital capacity. Additionally, respiratory muscles lose strength due to muscle atrophy and decreased fast-twitch fibers. These mechanisms can compromise ventilation, mucus clearance, and cough effectiveness, all essential for preventing bronchial congestion.

The effectiveness of Mechanical Insufflation-Exsufflation (MI-E) in airway clearance has been demonstrated in children and adults with neuromuscular pathologies.

Since the respiratory function of old people may be similar to that of patients with neuromuscular pathologies due to age-related loss of respiratory capacity and cough strength, it would be interesting to specifically study the use of MI-E in this population. Our previous study (ClinicalTrials.gov Identifier: NCT05090696) showed that old people tolerated MI-E well (low discomfort and no changes in vital signs). After the first session of bronchial clearance with MI-E, dyspnea decreased significantly (median Borg scale before session = 2.8 versus after = 1.8, p = 0.004). Additionally, cough strength increased across all sessions (mean pre = 130 vs. post = 145, p = 0.005).

Following this initial study, the investigators wondered if the use of MI-E would be more effective than a session of manual physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 or over, hospitalised in intensive care units or general medical wards, with bronchial congestion and a peak expiratory flow < 180 L/min, requiring respiratory physiotherapy
* Montreal Cognitive Assessment (MoCA) score ≥ 26
* Able to provide informed consent
* Affiliated with social health insurance

Exclusion Criteria:

* Neuromuscular disorders
* Spinal cord injury
* Contraindications to the use of mechanical insufflation-exsufflation:

  * History of bullous emphysema, surgical emphysema, or undrained pneumothorax
  * Recent barotrauma
  * Tracheoesophageal fistula
  * Bronchospasm
  * Hemodynamic instability
  * Refusal to participate.
* Inability to cough on command
* Pregnant or breastfeeding women
* People under protective legal measures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-09-18 (Estimated); Study Completion 2028-09-18 (Estimated)

PRIMARY OUTCOMES:
Variation in peak cough flow (PCF) | Day 1
  The variation in peak cough flow (PCF) is expressed as a percentage change from the pre-session value.
Variation in peak cough flow (PCF) | Day 2
  The variation in peak cough flow (PCF) is expressed as a percentage change from the pre-session value.

SECONDARY OUTCOMES:
Forced Vital Capacity | Day 1
  This outcomme will be assessed by an electronic spirometer. This value is in absolute values (LBTPS/sec) and as a percentage, taking into account the patient's age, sex and height.
Forced Vital Capacity | Day 2
  This outcomme will be assessed by an electronic spirometer. This value is in absolute values (LBTPS/sec) and as a percentage, taking into account the patient's age, sex and height.
Maximum Inspiratory and Expiratory Pressure | Day 1
  This outcome will be assess by an electronic spirometer in cmH2O
Maximum Inspiratory and Expiratory Pressure | Day 2
  This outcome will be assess by an electronic spirometer in cmH2O
Maximal Expiratory Volume in 1 second | Day 1
  This outcome will be assess by an electronic spirometer in percentage.
Maximal Expiratory Volume in 1 second | Day 2
  This outcome will be assess by an electronic spirometer in percentage.
Bronchial obstruction | Day 1
  This outcomme will be assess by an electronic spirometer with the Tiffenau index (Maximal expiratory volume in 1 second / Forced Vital Capacity).
Bronchial obstruction | Day 2
  This outcomme will be assess by an electronic spirometer with the Tiffenau index (Maximal expiratory volume in 1 second / Forced Vital Capacity).
Discomfort | Day 1
  Session discomfort using a numerical scale (0 - no discomfort; 10 - very uncomfortable session); session discomfort will be measured after each session.
Discomfort | Day 2
  Session discomfort using a numerical scale (0 - no discomfort; 10 - very uncomfortable session); session discomfort will be measured after each session.
Dyspnea | Up to day 2
  This using the modified Borg scale (0-no shortness of breath; 10-maximum shortness of breath felt during the session).

CONTACTS AND LOCATIONS:
Overall Officials: Claire Estenne, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (4):
- France (4):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - HCL Hôpital Edouard Herriot, Lyon
  - HCL Hôpital Louis Pradel, Lyon
  - Hôpital Saint Joseph Saint Luc, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estenne C, Dobija L, Pelletier-Visa M, Pereira B, Coudeyre E. Efficacy of using a mechanical insufflation-exsufflation versus manual respiratory physiotherapy on cough peak flow in hospitalised older adults in French hospitals: a protocol for a single-blind randomised clinical trial. BMJ Open. 2025 Oct 15;15(10):e105351. doi: 10.1136/bmjopen-2025-105351. PMID 41093324